CLINICAL TRIAL: NCT00219687
Title: Randomized Trial of Dispatcher-Assisted CPR:Chest Compression Alone Versus Chest Compression Plus Ventilation
Brief Title: Dispatcher-Assisted Resuscitation Trial (DART)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Public Health - Seattle and King County (Other Government)
Responsible Party: Principal Investigator, Susan Damon, Program Manager, Public Health - Seattle and King County
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RARC-0001-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Heart Arrest
Keywords: Heart arrest; Cardiopulmonary resuscitation; Dispatcher
MeSH Terms: conditions — Heart Arrest | interventions — Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): When a 911 call is determined to be a cardiac arrest, the caller reporting the event who needs or desires instructions to perform CPR while waiting for EMS to arrive will receive dispatcher-assisted CPR instructions with chest compressions only
  Interventions: Other: dispatcher-assisted CPR instructions with compressions only
- 2 (Active Comparator): When a 911 call is determined to be a cardiac arrest, the caller reporting the event who needs or desires instructions to perform CPR while waiting for EMS to arrive will receive dispatcher-assisted CPR instructions with chest compressions and breaths
  Interventions: Other: dispatcher-assisted CPR with compressions & ventilations

INTERVENTIONS:
Other: dispatcher-assisted CPR with compressions & ventilations — Delivery of telephone CPR instructions to lay callers with chest compressions and ventilations when the patient is identified to be in cardiac arrest
  Arms: 2
Other: dispatcher-assisted CPR instructions with compressions only — Delivery of telephone CPR instructions to lay callers with hands-only chest compressions when the patient is identified to be in cardiac arrest
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether dispatcher-assisted CPR instructions with compressions and ventilations versus dispatcher-assisted CPR instructions with compressions only improves survival from out-of-hospital cardiac arrests.

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest, a condition characterized by a person suddenly collapsing due to heart stoppage, is a leading cause of death in the United States. In out-of-hospital cardiac arrest, survival is dependent upon what the American Heart Association has termed the chain of survival which includes quick activation of the 9-1-1 system, prompt cardiopulmonary resuscitation (CPR), early defibrillation, and qualified advanced life support care (paramedic care). CPR allows for some circulation and delivery of oxygen to vital organs when the heart is no longer beating on its own. However, in some instances, the citizen bystander has not been trained in CPR, presenting a circumstance where the cardiac arrest victim may not receive CPR until the arrival of emergency medical services (EMS) personnel (i.e., paramedics). The delay in CPR adversely affects outcome and dcreases the chance of survival. In response to this need, the EMS Division of Public Health - Seattle and King County developed and instituted telephone CPR instructions that could be provided "on-the-spot" during a cardiac arrest by the emergency medical (9-1-1) dispatcher. The instructions are designed to be given over the phone to persons who have not had previous CPR training so that they can initiate CPR prior to the arrival of EMS personnel and have been termed "dispatcher-assisted" CPR. The dispatcher instructions provided by the dispatch agencies of King County include the standard "full" CPR protocol of ventilations (breathing into the victim's mouth to inflate the lungs) and chest compressions(pumping on the patients chest to help circulate the blood). The ventilations oxygenate the blood while the chest compressions pump the oxygenated blood forward. This EMS program has led to a considerable increase in the proportion of cardiac arrest victims in King County that receive citizen bystander CPR prior to EMS arrival and has been associated with improved survival (appendix 1).

Comparison: Dispatcher-assisted CPR instructions with compressions and ventillations compared to dispatcher-assisted CPR instructions with compressions only.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest events where CPR is not ongoing but a bystander is willing to attempt with assistance

Exclusion Criteria:

* Pregnancy
* Prisoners
* Cardiac arrest due to asphyxia, drowning, hanging, or electrocution

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5494 (Actual)
Dates: Start 2004-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Survival to hospital discharge | varied
  assessed at hospital discharge

SECONDARY OUTCOMES:
Neurological status at hospital discharge | varied
  assessed at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Rea, MD, MPH, Principal Investigator — Division of Emergency Medical Services, Public Health - Seattle and King County; Mickey S Eisenberg, MD, PhD, Principal Investigator — Division of Emergency Medical Services, Public Health - Seattle and King County
Locations (3):
- United States (2):
  - Thurston County Dispatch, Olympia, Washington
  - Division of Emergency Medical Services, Public Health - Seattle and King County, Seattle, Washington
- London Ambulance Service, London, England, United Kingdom

REFERENCES:
- [Derived] Rea TD, Fahrenbruch C, Culley L, Donohoe RT, Hambly C, Innes J, Bloomingdale M, Subido C, Romines S, Eisenberg MS. CPR with chest compression alone or with rescue breathing. N Engl J Med. 2010 Jul 29;363(5):423-33. doi: 10.1056/NEJMoa0908993. PMID 20818863